CLINICAL TRIAL: NCT05247190
Title: Treating Self-criticism in Adolescents: a Study With Single-case Experimental Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Östergötland (Other)
Responsible Party: Principal Investigator, Maria Zetterqvist, Ass professor, Region Östergötland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-04939
Record Dates: First submitted 2022-01-27; First posted 2022-02-18 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Adolescent - Emotional Problem; Adolescent Problem Behavior; Nonsuicidal Self Injury; Depressive Symptoms; Anxiety; Self-Criticism
Keywords: self-criticism; adolescents; group intervention; single-case experimental design
MeSH Terms: conditions — Self-Injurious Behavior; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Single-case experimental design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treating self-criticism (Experimental): 8-session group intervention targeting self-criticism given 2-hrs/week with booster session after 3-months.
  Interventions: Behavioral: Treating self-criticism

INTERVENTIONS:
Behavioral: Treating self-criticism — A psychological treatment given i a group format targeting self-criticism. The treatment is based on treatment principles from Cognitive behavior therapy, Self-compassion, Acceptance and Commitment Therapy and also contains psychoeducation. The group treatment consists of 8 sessions delivered once a week for 2 hrs during 8 weeks in a child- and adolescent psychiatric outpatient setting.

SUMMARY:
In this pilot study, the effect of a group intervention targeting self-criticism in adolescents in a clinical child- and adolescent psychiatric outpatient setting will be examined using a single-case experimental design (AB). Participants will be randomized to multiple baseline with weekly measures. Our primary outcomes, measured weekly, are self-criticism, nonsuicidal self-injury and symptoms of depression and anxiety, as well as an individually chosen behavior driven by self-criticism. Secondary outcomes are self-compassion, psychological flexibility, quality of life and functioning. In addition to the weekly administered questionnaires, before and after measures, and 3- and 6-month follow-up will be collected. After the treatment, participants will also be interviewed about their experiences of targeting self-criticism.

ELIGIBILITY:
Inclusion Criteria:

* Patient at the child- and adolescent psychiatric clinic in Linköping, Sweden.
* 15 to 18 years
* an adequate understanding of the Swedish language
* cognitively capable of giving informed consent
* scoring 26 or above on subscale "Inadequate self" and 8.5 or above on subscale "Hated Self" on questionnaire Forms of Self-Criticism and Self-Reassuring Scale (FSCRS)
* the treatment is transdiagnostic so all diagnoses are included (See exclusion criteria for exceptions).

Exclusion Criteria:

* severe anorexia, BMI ≤ 16
* ongoing substance abuse
* diagnosed intellectual disability
* needing interpreter for translation of Swedish language
* participants who cannot give informed consent

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Self-criticism | Change from baseline (phase A) at intervention (phase B) 8 weeks, and at 3- and 6- months
  Forms of Self-Criticism and Self-Reassuring Scale (FSCRS; Gilbert et al., 2004)

SECONDARY OUTCOMES:
Self-Compassion | Change from before to after intervention, and at 3- and 6- month follow-up
  Self-Compassion Scale, short form (SCS; Raes et al., 2011)
Psychological flexibility | Change from before to after intervention, and at 3- and 6- month follow-up
  Avoidance and Fusion Questionnaire for Youth (AFQ-Y8; Greco et al., 2008).
Quality of life and functioning | Change from before to after intervention, and at 3- and 6- month follow-up
  The Work and Social Adjustment Scale, youth version (WSAS-Y; Mundt et al., 2002).
Symptoms of depression | Change from baseline (phase A) at intervention (phase B) 8 weeks, and at 3- and 6- months
  Montgomery Åsberg Depression Rating Scale, self-report version (MADRS-S; Montgomery et al., 1979).
Symptoms of anxiety | Change from baseline (phase A) at intervention (phase B) 8 weeks, and at 3- and 6- months
  Liebowitz Social Anxiety Scale, self-report (LSAS; Liebowitz, 1987)
Nonsuicidal self-injury | Change from baseline (phase A) at intervention (phase B) 8 weeks, and at 3- and 6- months
  Selected items from Self-Injurious Thoughts and Behaviors interview (SITBI; Nock et al., 2007), Deliberate self-harm inventory (DSHI; Gratz et al., 2001) och Clinician Administered Nonsuicidal self-injury Disorder Interview (CANDI; Gratz et al., 2015)
Individually chosen behavior | Change from baseline (phase A) at intervention (phase B) 8 weeks, and at 3- and 6- months
  A behavior driven by self-criticism

CONTACTS AND LOCATIONS:
Overall Officials: Maria Zetterqvist, PhD, Principal Investigator — Region Östergötland and Linköping university
Locations (1):
- Region Ostergotland BUP-kliniken, Linköping, Sweden